CLINICAL TRIAL: NCT02188797
Title: Brief AOD Use and Sexual Risk Reduction Group MI Intervention for Homeless
Brief Title: Substance Use and Sexual Risk Reduction Intervention for Homeless Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA034813 (NIH)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Substance Use; Sexual Risk Behavior
Keywords: homeless; young adults; substance use; HIV risk; sexual risk behavior; group motivational interviewing
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group MI risk reduction program (Experimental): Participants receive four 1-hour group motivational interviewing sessions focused on reducing substance use and sexual risk behavior. They also receive an HIV information brochure and Community Resource Guide.
  Interventions: Behavioral: Group MI risk reduction program
- Usual care control (No Intervention): Participant receive HIV information brochure and Community Resource Guide.

INTERVENTIONS:
Behavioral: Group MI risk reduction program
  Arms: Group MI risk reduction program

SUMMARY:
The goal of this study is to evaluate a group-based motivational interviewing (MI)-delivered risk reduction program for homeless young adults. It is hypothesized that youth who participate in the program will show greater reductions in substance use intentions, behavior and consequences, as well as sexual activity intentions and risk behavior, over a 3-month period compared to a usual care control sample of youth who do not participate in the program.

DETAILED DESCRIPTION:
This study addresses an important gap in prevention services for homeless youth by conducting a pilot test of an innovative 4-session integrated substance use and sexual risk reduction program for this population that is feasible to deliver in settings where these youth seek services. The study has 2 specific aims:

Aim 1: Investigate whether homeless youth who participate in the program show reductions in substance use and intentions, behavior and consequences, as well as sexual activity intentions and risk behavior, over a 3-month period compared to a usual care control sample of youth who do not receive the program.

Aim 2: Gain a better understanding of intervention effects by exploring whether improvements in self-efficacy, readiness to change, outcome expectancies, and exposure to peer substance use and offers serve as explanatory mechanisms for reductions in substance use- and sexual activity- related intentions and risk behaviors among youth who participate in the program.

The program will be evaluated using a form of group-randomized design, although with crossover of conditions and groups to avoid the problems of power reduction associated with conventional group randomization. The unit of analysis will be the individual, but individuals will be assigned to groups based on the agency where they are seeking services. Youth at two drop-in centers serving homeless youth will either be in the intervention condition or a "usual care" control condition. The field period will be divided into four phases. The two agencies will alternate across phases in serving as the "intervention site" or "control site," with each agency having a total of two intervention phases and two control phases.

Intervention Condition: This condition involves a four-session voluntary intervention that is delivered within a drop-in center setting and is based on the investigator's previous intervention work with adolescents and young adults. Each session lasts approximately 1 hour. The intervention focuses on both sexual risk behavior and substance use. Although some sessions focus more heavily on sexual risk and others on substance use, each session includes content that emphasizes the interrelated nature of these two risk behaviors. In all sessions, participants will receive a personalized feedback sheet that specifically addresses a topic being discussed during that particular session. An motivational interviewing approach will be used to present material during the group sessions.

"Usual Care" Condition: The "usual care" condition reflects the resources typically available in settings that serve homeless youth: an HIV informational brochure that discusses the connection between substance use and HIV risk, and a Community Resource Guide that lists free or low-cost substance use and HIV-related services.

ELIGIBILITY:
Inclusion Criteria:

* between 18-24 years, receiving services at one of the participating drop-in centers, planning to be in the study area for the next month

Exclusion Criteria:

* obvious cognitive impairment observed during screening process; non-English speaking

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in substance use | baseline, 3 months
  past month quantity-frequency of alcohol and marijuana; past 3 months frequency of alcohol, binge drinking, marijuana, crack, cocaine, heroin, methamphetamine, ecstasy, hallucinogens, inhalants, prescription drug misuse
Change in substance use intentions | baseline, 3 months
  Intentions to use the following in the next 3 months: alcohol; marijuana; other drugs
Change in negative consequences from drinking | baseline, 3 months
Change in use of drinking protective strategies | baseline, 3 months
Change in number of different sex partners | baseline, 3 months
Change in condom use | baseline, 3 months
Change in substance use before or during sex | baseline, 3 months
Change in HIV knowledge | baseline, 3 months
Change in sex-related protective strategies | baseline, 3 months
Change in sexual intentions | baseline, 3 months
  Separate items for intentions for buying/getting condoms, carrying condoms, talking to partner about condoms, using condoms, using condoms when drinking or using drugs, getting tested
Change in HIV testing | baseline, 3 months
  Self-report of being tested in lifetime, past 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - My Friend's Place, Hollywood, California
  - Safe Place for Youth, Venice Beach, California